CLINICAL TRIAL: NCT03239756
Title: Phase 1 Trial of a Fully Human Monoclonal Antibody of Receptor Activator for Nuclear Factor-κ B Ligand (RNAKL, TK006) Safety, Pharmacokinetics, and Pharmacodynamics in Patients With Breast Cancer-related Bone Metastases
Brief Title: Assessment of TK006 in Patients With Breast Cancer-related Bone Metastases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-TK006-102
Record Dates: First submitted 2017-07-28; First posted 2017-08-04 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 60 mg single dose cohort (Experimental): patients would receive a 60 mg single dose of TK006.
  Interventions: Biological: TK006
- 120 mg single dose cohort (Experimental): patients would receive a 120 mg single dose of TK006.
  Interventions: Biological: TK006
- 180 mg single dose cohort (Experimental): patients would receive a 180 mg single dose of TK006.
  Interventions: Biological: TK006
- 120 mg Q4W cohort (Experimental): patients would receive 120 mg TK006 every 4 weeks, for a total of 3 doses.
  Interventions: Biological: TK006

INTERVENTIONS:
Biological: TK006 — Subcutaneous injection
  Other Names: fully human monoclonal anti-RANKL antibody

SUMMARY:
This is a single-center, open-label, dose-escalating study to evaluate the safety, pharmacokinetics, immunogenicity, and preliminary efficacy of single and multiple subcutaneous injection TK006 in patients with breast cancer-related bone metastases.

DETAILED DESCRIPTION:
This is an single-center, open-label, dose-escalating study to evaluate the safety, pharmacokinetics, immunogenicity, and preliminary efficacy of single and multiple subcutaneous injection TK006 in patients with breast cancer-related bone metastases. It contains 4 cohorts：60 mg single-dose conhort, 120 mg single-dose conhort, 180 mg single-dose conhort and 120 mg Q4W （one dose every 4 weeks, 3 dose totally） conhort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients provide written informed consent voluntarily；
2. 18~65 years old；
3. Patients with pathology confirmed breast cancer radiological evidence with bone metastasis；
4. Eastern Cooperative Oncology Group(ECOG) performance status≤2
5. Anticipated life span≥6-month；
6. Adequate reservation of hematopoiesis, liver and kidney functions:

   * Absolute neutrophil count (ANC) ≥1.5×10^9/L
   * Absolute platelet count (PLT) ≥100×10^9/L
   * Hemoglobin (Hb) ≥90 g/L
   * Total bilirubin (TBIL) ≤1.0 time the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.0 ULN
   * Serum creatinine (sCr) ≤2.0 ULN
7. Albumin-adjusted calcium≥2.0 mmol/L, ≤2.9 mmol/ L(Calcium supplements are not allowed within 8 hours before examination).

Exclusion Criteria:

1. Hypersensitivity to any investigational medicine or supplements in this study.
2. Women in Pregnancy or nursing.
3. Anti-human immunodeficiency virus (HIV) antibody positive.
4. Patients with hepatitis B virus DNA ≥10^5 copies/mL or active hepatitis C would not be selected. Stable hepatitis B or hepatitis C defined as AST/ALT≤2 ULN will not be selected as well if patients are not treated with antiviral therapy while receving immunosuppressive therapy or chemotherapy meanwhile.
5. Prior malignancies (excluding the targeted breast cancer, basal cell carcinoma, or cervical cancer in situ) within 3 years.
6. Uncontrolled systemic diseases, or organic or mental disorders that could affect compliance.
7. Central nervous system metastasis that is symptomatic or require treatment.
8. Unresolved toxicities ≥2 grades from previous chemo-therapy (excluding alopecia).
9. Major surgery of bone or trauma within 4 weeks before the first dosing.
10. Fracture of long bone within 90-day before the first dosing.
11. Radiation therapy to bone within 2 weeks or treatment with radioisotopes within 8 weeks before the first dosing.
12. Treatment with diphosphonate within 30-day or administration of calcitonin, parathyroid hormone-related peptides, mithramycin, gallium nitrate or strontium ranelate within 6-month before the first dosing. Plan to receive systemic treatment with glucocorticosteroids over a long period during the trial.
13. Hyperthyroidism or hypothyroidism, unless hypothyroidism patients are receiving regular treatment with thyroid hormone and:

1) Thyroid stimulating hormone (TSH) is normal, or 2) TSH>4.78μIU/Ml, ≤10.0μIU/mL and thyroxine (T4) is normal. 14. Disorders of hypoparathyroidism or hyperparathyroidism, osteomalacia, rheumatoid arthritis, acute attack of osteoarthritis, gout, Paget's disease, malabsorption syndrome, ascites, or other diseases that could affect bone metabolism.

15. Previous or existing osteomyelitis or osteonecrosis of jaw, odontia or jaw diseases which are in active or require invasive operations, unhealing wound of oral surgery, or planned invasive dental operations during this trial.

16. Has been selected for the study of other test devices or test drugs, or the duration of the clinical studies that have taken less than 30 days or 5 half-lives or biological effects, whichever is longer.

17. Other situations which are not suitable for participation judged by the principal investigator (PI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) which are related to TK006 assessed by CTCAE v4.03 | single dose cohort：112 days, multiple dose cohort：140 days
  Collect the information of AEs and SAEs, vital sign, physical examination, laboratory examination and electrocardiogram during the trial.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to time 'last' where last is the last time point after administration [AUClast] | single dose cohort：112 days, multiple dose cohort：140 days
  Calculated by the linear trapezoidal method.
Area under the plasma concentration-time curve from time zero to infinity [AUC0-inf] | single dose cohort：112 days, multiple dose cohort：140 days
  Calculated by the linear trapezoidal and extrapolation method.
Maximum observed maximum plasma concentration [Cmax] | single dose cohort：112 days, multiple dose cohort：140 days
  The maximum (or peak) serum concentration that TK006 achieves after the drug has been administrated and before the administration of a second dose.
Time to reach the maximum observed plasma concentration [Tmax] | single dose cohort：112 days, multiple dose cohort：140 days
  The time at which the Cmax is observed.
Terminal elimination half-life[T1/2] | single dose cohort：112 days, multiple dose cohort：140 days
  The time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose.
bioavailability corrected apparent volume of the central compartment cleared of drug per unit [Cl/F] | single dose cohort：112 days, multiple dose cohort：140 days
  The apparent volume of the central compartment cleared of drug per unit time was estimated using the formula: Cl/F = Dose / AUC0-∞
bioavailability corrected apparent volume of distribution [Vd/F] | single dose cohort：112 days, multiple dose cohort：140 days
  Apparent volume of distribution based on the terminal elimination phase.
urine creatinine corrected cross-linked N-telopeptides of type I collagen [uNTX/Cr] | single dose cohort：112 days, multiple dose cohort：140 days
  For singel dose cohort, detecting the level of uNTX at screening period, day 0 (before dosing)、day 1, day 7, day 14, day 28, day 56, day 84 and day 112 For multiple dose cohort：detecting the level of uNTX at screening period, day 0 (before dosing)、day 1, day 7, day 14, day 28 (before dosing), day 56 (before dosing), day 84 and day 140.
  Assessing the change of uNTX level to baseline and the uNTX should be corrected by urine creatinine.
serum bone alkaline phosphatase [bALP] | single dose cohort：112 days, multiple dose cohort：140 days
  Assessing the change of serum bALP level to baseline. For singel dose cohort, detecting the level of uNTX at screening period, day 0 (before dosing)、day 1, day 7, day 14, day 28, day 56, day 84 and day 112 For multiple dose cohort：detecting the level of uNTX at screening period, day 0 (before dosing)、day 1, day 7, day 14, day 28 (before dosing), day 56 (before dosing), day 84 and day 140.
anti-drug antibody [ADA] | single dose cohort：112 days, multiple dose cohort：140 days
  Quantitative assay the ADA. For single cohort, the ADA titer would be detected at day 0 (before dosing) and day 56.
  For multiple dose cohort, the ADA titer would be detected at day 0 (before dosing), day 28 (before dosing), day 56 (before dosing), day 84 and day 140.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang H Y, Study Director — Jiangsu T-Mab Biopharma Co.,Ltd
Locations (1):
- the first affiliated hospital with Nanjing University, Nanjing, Jiangsu, China